CLINICAL TRIAL: NCT04884009
Title: An Open-label, Multicenter PhaseⅡ Study of SHR-1701 in Combination With or Without Famitinib Malate for the Treatment of Extensive Stage Small Cell Lung Cancer After Previous Systemic Chemotherapy Failure
Brief Title: A Trial of SHR-1701 in Combination With and Without Famitinib Malate in Patients With Extensive Stage Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1701-II-209
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — SHR-1701

STUDY DESIGN:
Intervention Model Description: SHR-1701 in combination with or without famitinib
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1701+ Famitinib (Experimental)
  Interventions: Drug: SHR-1701； Famitinib
- SHR-1701 (Experimental)
  Interventions: Drug: SHR-1701

INTERVENTIONS:
Drug: SHR-1701； Famitinib — SHR-1701+ Famitinib
  Arms: SHR-1701+ Famitinib
Drug: SHR-1701 — SHR-1701
  Arms: SHR-1701

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of SHR-1701 in combination with or without famitinib malate for the treatment of extensive stage small cell lung cancer after the failure of previous systemic chemotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participated in the clinical study, understood the study procedures and are able to sign the informed consent form.
2. 18 to 75 years old, male or female.
3. Histologically or cytologically confirmed extensive stage small cell lung cancer（ED-SCLC）.
4. ECOG Performance Status of 0 or 1.
5. Adequate hematological, hepatic and renal function.
6. Female subjects of child-bearing potential must have a negative serum HCG test before treatment.

Exclusion Criteria:

1. Histologically or cytologically confirmed mixed SCLC and NSCLC.
2. Untreated central nervous system metastases.
3. Cancerous meningitis (meningeal metastasis).
4. Uncontrolled pleural effusion, pericardial effusion or ascites.
5. Tumor infiltration into the great vessels on imaging;
6. Hemoptysis symptoms and maximum daily hemoptysis ≥ 2.5ml occurred within 1 month.
7. Uncontrolled tumor-related pain.
8. Malignancies other than SCLC within 5 years.
9. Systemic antitumor therapy was received 4 weeks prior to trial treatment.
10. History of autoimmune diseases.
11. Significant cardiovascular disease.
12. Inadequately controlled hypertension.
13. Known history of testing positive test for HIV or known AIDS.
14. Patients with active hepatitis B or hepatitis C
15. Severe infections within 4 weeks prior to trial treatment.
16. Active tuberculosis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2021-05-31 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) based on RECIST 1.1 criteria | up to approximately 1 year.

SECONDARY OUTCOMES:
Progression free survival (PFS) based on RECIST 1.1 criteria | up to approximately 1 year.
Disease control rate (DCR) based on RECIST 1.1 criteria | up to approximately 1 year.
Duration of response (DoR) | up to approximately 1 year
Overall survival (OS) | up to approximately 1 year
AEs+ SAEs determined by NCI-CTCAE V5.0 | Baseline until up to 90 days after end of treatment.